CLINICAL TRIAL: NCT03520374
Title: Evaluating the Effectiveness of a Self-instructional Ultrasound Training Program at Teaching Aspiration Risk Assessment Through Gastric Ultrasound
Brief Title: Bedside Ultrasound of Gastric Contents in Pediatric Populations
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Chi-Ho Ban Tsui, Principal Investigator, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 44959
Record Dates: First submitted 2018-04-27; First posted 2018-05-09 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Gastric Contents
Keywords: ultrasound; gastric contents
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Healthy adult volunteers (Other): Novice ultrasonographers will be taught to assess gastric contents with a short and simple educational program. Each novice will assess the gastric contents of 3 healthy adult volunteers using the clinical algorithm for gastric ultrasound and aspiration risk assessment - giving an antral grade for each subject (a score of 0-2). Each novice ultrasound assessment will be video recorded. In the weeks following this evaluation, expert ultrasonographers will observe each video and give their own scores for each subject using the antral grading system.
  Interventions: Diagnostic Test: Ultrasonography
- Pediatric patients (Other): Novice ultrasonographers will be taught to assess gastric contents with a short and simple educational program. Each novice will assess the gastric contents of 3 pediatric patients undergoing surgery in the preoperative area or the in-patient unit using the clinical algorithm for gastric ultrasound and aspiration risk assessment - giving an antral grade for each subject (a score of 0-2). Each novice ultrasound assessment will be video recorded. In the weeks following this evaluation, expert ultrasonographers will observe each video and give their own scores for each subject using the antral grading system.
  Interventions: Diagnostic Test: Ultrasonography

INTERVENTIONS:
Diagnostic Test: Ultrasonography — Ultrasonography use for the evaluation of gastric contents

SUMMARY:
Perioperative aspiration of gastric contents is a rare but serious adverse event. The risk of aspiration can be estimated by perioperative evaluation of stomach contents with ultrasound using a validated technique and scoring system. A lack of knowledge or familiarity is frequently cited by anesthesia providers as a rationale for not performing perioperative ultrasound assessments. The purpose of this study is to determine whether novice ultrasonography users (medical students, undergraduates, or inexperienced anesthesiologists) can be effectively taught a technique to evaluate stomach contents as compared to experts in ultrasonography.

DETAILED DESCRIPTION:
This study will be conducted in two arms. For part 1, we will evaluate the efficacy of the self-taught course at producing accurate reads among novice ultrasound users on ideal, cooperative, adult subjects. For part 2, we will evaluate the effectiveness of the course through an identical study that uses clinical pediatric patients as subjects.

Using available literature and established standards for gastric ultrasound, a 15-minute ultrasound training video course will be designed that gives instruction on ultrasound orientation, use, and the antral scoring system of gastric contents. Ten novice ultrasound users will be selected by study personnel on a volunteer basis from a pool of undergraduate students, medical students, and inexperienced anesthesiologists acting as research interns.

For Part 1, 30 healthy adult volunteers with unknown gastric-content status will be recruited to serve as scanning subjects. For Part 2 (which will only begin after successful completion of Part 1), 30 patients will be recruited from pediatric hospital populations undergoing surgery in the preoperative area or the in- patient unit.

Each novice will assess the gastric contents of 6 subjects (3 in Part 1 and 3 in Part 2) using the clinical algorithm for gastric ultrasound and aspiration risk assessment - giving an antral grade for each subject (a score of 0-2). Each novice ultrasound assessment will be video recorded. In the weeks following this evaluation, expert ultrasonographers will observe each video and give their own scores for each subject using the antral grading system.

ELIGIBILITY:
Inclusion Criteria:

Patients must:

1. be between ages of 2-60 years of age
2. have parental consent for children 2-17 years of age, or if the participant is 18 years or older, the participant must sign the ICF for them self as an adult
3. undergoing interventional radiology procedures under general anesthesia or located at an inpatient/outpatient facility at LPCH if they are a pediatric patient
4. must be over 18 years of age if a healthy volunteer

Exclusion Criteria:

1. Patients undergoing emergent surgical procedures
2. BMI greater than 24

Ages: 2 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-08-02 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Novice vs Expert Ultrasonographers Gastric Evaluation | Novice ultrasonographers: for pediatric patients - after anesthesia induction and before the procedure start, for healthy volunteers - hours following signing the consent form. Expert ultrasonographers: weeks following the initial evaluation by novices.
  The gastric evaluation of novice and expert ultrasonographers will be compared based on a 3-point numerical evaluation.

SECONDARY OUTCOMES:
Time elapsed to reach gastric evaluation | Novice ultrasonographers: for pediatric patients - after anesthesia induction and before the procedure start, for healthy volunteers - hours following signing the consent form. Expert ultrasonographers: weeks following the initial evaluation by novices.
  Time elapsed to reach gastric evaluation will be assessed in both novice and expert ultrasonographers

CONTACTS AND LOCATIONS:
Overall Officials: Ban CH Tsui, MD, Study Director — Stanford University
Locations (1):
- LPCH/SHC, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No
All data will be de-identified. Data will be used collectively for research analysis.

REFERENCES:
- [Result] Arzola C, Perlas A, Siddiqui NT, Downey K, Ye XY, Carvalho JCA. Gastric ultrasound in the third trimester of pregnancy: a randomised controlled trial to develop a predictive model of volume assessment. Anaesthesia. 2018 Mar;73(3):295-303. doi: 10.1111/anae.14131. Epub 2017 Dec 19. PMID 29265187
- [Result] Spencer AO, Walker AM, Lardner DR, Perlas A. Reply to Schmitz et al. regarding 'Ultrasound assessment of gastric volume in the fasted pediatric patient undergoing upper gastrointestinal endoscopy: development of a predictive model using endoscopically suctioned volumes'. Paediatr Anaesth. 2016 Jun;26(6):672-3. doi: 10.1111/pan.12915. No abstract available. PMID 27119308
- [Result] Kruisselbrink R, Arzola C, Endersby R, Tse C, Chan V, Perlas A. Intra- and interrater reliability of ultrasound assessment of gastric volume. Anesthesiology. 2014 Jul;121(1):46-51. doi: 10.1097/ALN.0000000000000193. PMID 24595113
- [Result] Khurana J, Gartner SC, Naik L, Tsui BCH. Ultrasound Identification of Diaphragm by Novices Using ABCDE Technique. Reg Anesth Pain Med. 2018 Feb;43(2):161-165. doi: 10.1097/AAP.0000000000000718. PMID 29315130